CLINICAL TRIAL: NCT02794428
Title: Targeted Chemoprevention of Gastric Carcinogenesis in High Risk Populations
Brief Title: Chemoprevention of Gastric Carcinogenesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Prevention Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas Morgan, Director, Latin America sites, Vanderbilt Institute for Global Health, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: VICC GI 1527; 6R01CA190612-03 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-06-09 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer; Gastric Intestinal Metaplasia
Keywords: Gastric adenocarcinoma; Gastric intestinal metaplasia; Atrophic gastritis; Gastric premalignant lesion
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Eflornithine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eflornithine (Active Comparator)
  Interventions: Drug: Eflornithine
- Eflornithine Placebo (Placebo Comparator)
  Interventions: Other: Eflornithine placebo

INTERVENTIONS:
Drug: Eflornithine — Eflornithine*, 2 tablets, Oral, Daily for 18 months
  Arms: Eflornithine
Other: Eflornithine placebo — Eflornithine placebo, 2 tablets, Oral, Daily for 18 months
  Arms: Eflornithine Placebo

SUMMARY:
A clinical study of the efficacy of oral alpha-difluoromethylornithine (eflornithine or DFMO) in male and female subjects ages 30-60 with gastric premalignant lesions in two high risk regions of Latin America.

DETAILED DESCRIPTION:
Primary Objective

- The difference in cell DNA damage between patients treated with DFMO and patients treated with placebo at 6 months. The cell DNA damage is measured using the percent positive gastric epithelial cells assessed by IHC for gamma H2AX. The mean difference between the two groups at 6 months will be calculated, accounting for their baseline measurements.

Secondary Objectives

* The difference in cell DNA damage between patients treated with DFMO and patients treated with placebo for 18 months, and then followed for an additional 6 months. The cell DNA damage is measured using the percent positive gastric epithelial cells assessed by IHC for gamma H2AX. The mean difference between the two groups at 18 and 24 months will be calculated, accounting for their baseline measurements.
* The differences in the gastritis histopathology score between patients treated with DFMO and patients treated with placebo for a total of 18 months, and followed for an additional 6 months. The gastritis histopathology score is measured with a quantitative scale 0.0-6.0, for atrophy, intestinal metaplasia, and dysplasia. The mean differences between the two groups at 6, 18, and 24 months will be calculated using mixed models, accounting for their baseline measurements.
* Number of patients with quantitative toxicities. Toxicities will be assessed per CTCAE criteria, and each toxicity will be assigned an adverse event (AE) term according to CTCAE definitions (each AE term = unique representation of a specific event used for medical documentation and scientific analyses), and graded as defined by CTCAE (grade 1 = mild; grade 2 = moderate; grade 3 = severe or significant but not immediately life-threatening; grade 4 = life-threatening; grade 5 = death).
* To evaluate whether candidate single nucleotide polymorphisms (SNPs) relevant to eflornithine (DFMO) efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of a premalignant lesion of the stomach, atrophic gastritis or intestinal metaplasia
* Patients must have a pure tone audiometry evaluation to document air conduction within 60 days prior to randomization.
* Patients must have adequate blood counts as evidenced by the following results (obtained within 60 days):

  * Blood counts: WBC ≥4.0 /mcL, platelets ≥100,000 /mcL and hemoglobin ≥11.0 g/dL
  * Kidney function: Creatinine <1.6 x IULN (institutional upper limit of normal)
  * Liver function tests: Bilirubin ≤2.0 mg/dL and AST (SGOT) or ALT (SGPT) ≤2 x IULN

Exclusion Criteria:

* Subjects with dysplasia (indeterminate, low grade, high grade) are not eligible for participation
* Patients must not have a significant medical or psychiatric condition that would preclude study completion.
* Patients with hearing loss ≥30 dB in any of the tested frequencies (250 Hz, 500 Hz, 1,000 Hz, 2,000 Hz, 4,000 Hz, 8,000 Hz) are not eligible.
* Patients must not have known hypersensitivity to eflornithine or the excipients.
* Patients must not be receiving corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or anticoagulants on a regular or intermittent basis.
* Patients must not have a significant cardiovascular disease history, including uncontrolled blood pressure (sBP > 150 mmHg), myocardial infarction, cerebrovascular accident, or heart failure (New York Heart Association Class III, or IV).
* Patients must not have a history of gastric or esophageal cancer, gastric resection or surgery, peptic ulcer disease (within 6 months), H. pylori treatment (within 6 months), or inflammatory bowel disease.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for >5 years.
* Patients must not be receiving corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or anticoagulants on a regular or intermittent basis.
* Patients must not be pregnant or nursing (due to eflornithine pregnancy class C). Women and men of reproductive potential must have agreed to use an effective contraceptive method.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Morgan, MD, Study Chair — Vanderbilt University Medical Center, Vanderbilt-Ingram Cancer enter; Keith Wilson, MD, Principal Investigator — Vanderbilt University Medical Center, Vanderbilt-Ingram Cancer enter
Locations (2):
- Ministry of Health, Hospital de Occidente, Copán, Honduras
- University of Puerto Rico, Comprehensive Cancer Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Period: 6 Months (Primary End Point)
Arm/Group | Eflornithine | Eflornithine Placebo
Started | 45 | 46
Completed | 36 | 42
Not Completed | 9 | 4
Period: 18 Months (Secondary Endpoint)
Arm/Group | Eflornithine | Eflornithine Placebo
Started | 36 | 42
Completed | 31 | 38
Not Completed | 5 | 4
Period: 24 Months (End of Study)
Arm/Group | Eflornithine | Eflornithine Placebo
Started | 31 | 38
Completed | 26 | 29
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eflornithine | Eflornithine Placebo | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 46 | 91
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 45 | 46 | 91
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2 | 3 | 5
  Honduras | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Cell DNA Damage, Based on Percent Positive Cells, Between Patients Treated With DFMO and Patients Treated With Placebo at 6 Months.
Description: The cell DNA damage is measured using the percent positive gastric epithelial cells assessed by IHC for gamma H2AX.The mean difference between the two groups at 6 months will be calculated, accounting for their baseline measurements.
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: Percentage of positive cells
Arm/Group | Eflornithine | Eflornithine Placebo
Number analyzed (Participants) | 32 | 37
Percentage of positive cells | 5.07 (21.05) | 7.32 (21.60)

2. Secondary Outcome: The Difference in Cell DNA Damage Between Patients Treated With DFMO and Patients Treated With Placebo for 18 Months, and Then Followed for an Additional 6 Months.
Description: The cell DNA damage is measured using the percent positive gastric epithelial cells assessed by IHC for gamma H2AX. The mean difference between the two groups at 18 and 24 months will be calculated, accounting for their baseline measurements.
Time Frame: at 18 and 24 months
Reporting Status: Not Posted, anticipated posting 2025-05

3. Secondary Outcome: The Differences in the Gastritis Histopathology Score Between Patients Treated With DFMO and Patients Treated With Placebo for a Total of 18 Months, and Followed for an Additional 6 Months.
Description: The gastritis histopathology score is measured with a quantitative scale 0.0-6.0, for atrophy, intestinal metaplasia, and dysplasia. The mean differences between the two groups at 6, 18, and 24 months will be calculated using mixed models, accounting for their baseline measurements.
Time Frame: at 6, 18 and 24 months
Reporting Status: Not Posted, anticipated posting 2025-05

4. Secondary Outcome: Number of Patients With Quantitative Toxicities.
Description: Toxicities will be assessed per CTCAE criteria, and each toxicity will be assigned an adverse event (AE) term according to CTCAE definitions (each AE term = unique representation of a specific event used for medical documentation and scientific analyses), and graded as defined by CTCAE (grade 1 = mild; grade 2 = moderate; grade 3 = severe or significant but not immediately life-threatening; grade 4 = life-threatening; grade 5 = death).
Time Frame: at 6, 18, and 24 months
Reporting Status: Not Posted, anticipated posting 2025-05

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Eflornithine | Eflornithine Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/45 | 2/46
Other Adverse Events (participants affected / at risk) | 2/45 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eflornithine (N=45) | Eflornithine Placebo (N=46)
Hypertensive urgency (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eflornithine (N=45) | Eflornithine Placebo (N=46)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02794428/Prot_SAP_000.pdf